CLINICAL TRIAL: NCT00002016
Title: A Phase I/II Trial to Assess the Safety and Tolerance of Escalating Doses of a Human Anti-Cytomegalovirus Monoclonal Antibody (SDZ MSL-109) in Patients With the Acquired Immunodeficiency Syndrome and CMV Retinitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 071B; Study No B103
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1993-04

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Retinitis; Ganciclovir; Cytomegalovirus; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome; Antibodies, Monoclonal
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Retinitis; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome | interventions — sevirumab

INTERVENTIONS:
Drug: Sevirumab

SUMMARY:
To determine the safety and tolerance of 3 dosage levels of human anti-cytomegalovirus (CMV) monoclonal antibody (SDZ MSL-109) when administered once every 2 weeks for a total of 8 doses during the maintenance phase of ganciclovir (DHPG) therapy to patients with AIDS and documented evidence of CMV retinitis. In addition for those patients with positive CMV cultures upon entry into this trial a preliminary attempt will be made to assess the potential in vivo antiviral effects of the concomitant administration of DHPG and SDZ MSL-109.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Zidovudine (AZT) < 600 mg/day.
* Experimental maintenance or prophylactic therapy with an approved therapeutic agent for a non-viral opportunistic infection.
* Trimethoprim / sulfamethoxazole (TMP / SMX).
* Pyrimethamine / sulfadoxine.
* Aerosolized pentamidine.
* Ketoconazole.
* Flucytosine (5-FC).
* Antituberculosis therapy.

Concurrent Treatment:

Allowed:

* Maintenance phase of ganciclovir (DHPG) therapy.

Patients must have:

* AIDS with documented ophthalmologic findings consistent with cytomegalovirus (CMV) retinitis whose retinal lesions are less than 750 microns from the fovea and who have visual symptoms of CMV retinitis.
* Completed the treatment induction phase with ganciclovir (DHPG) and be about to participate in the maintenance phase DHPG therapy.
* Expected survival of = or > 6 months.
* Willingness and ability to give written informed consent. A copy of the signed and witnessed consent form must be maintained with the investigator's study files.
* Seropositive for the presence of circulating anti-CMV immunoglobulin.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Significant pulmonary dysfunction.
* Uncontrolled or unstable diabetes.
* Significant cardiovascular disease including uncontrolled hypertension, congestive heart failure, cardiac arrhythmia, angina pectoris, or a history of myocardial infarction within one year of entry into the study.
* Coagulation or hemorrhagic disorders.
* Any active severe opportunistic infection.

Concurrent Medication:

Excluded:

* Therapy with amphotericin B or fluconazole.
* Any other investigational drug.
* Biologicals including immunoglobulin therapy, granulocyte-macrophage-colony-stimulating-factor (GM-CSF), erythropoietin alpha, or any interleukin.

Patients with the following are excluded:

* Any significant organ system dysfunction as described in Exclusion Co-existing Conditions.
* Any other severe concomitant clinical condition.

Prior Medication:

Excluded within 2 weeks of study entry:

* Therapy with amphotericin B or fluconazole.
* Any other investigational drug.
* Biologicals including immunoglobulin therapy, granulocyte-macrophage-colony-stimulating factor (GM-CSF), erythropoietin alpha, or any interleukin.
* Excluded:
* Prior treatment with monoclonal antibodies derived from any animal species.

Prior Treatment:

Excluded within 2 weeks of study entry:

* Major surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Univ TX Galveston Med Branch, Galveston, Texas

REFERENCES:
- [Background] Tolpin M, Pollard R, Tierney M, Nokta M, Wood D, Hirsch M. Combination therapy of cytomegalovirus (CMV) retinitis with a human monoclonal anti-CMV antibody (SDZ MSL 109) and either ganciclovir (DHPG) or foscarnet (PFA). Int Conf AIDS. 1993 Jun 6-11;9(1):54 (abstract no WS-B11-2)